CLINICAL TRIAL: NCT04838093
Title: COVID-19 Testing in Patients With Vascular Disorders - a Prospective Cohort Study at a Tertiary Care Hospital
Brief Title: COVID-19 Testing in Patients With Vascular Disorders
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Mohammad M. Kasiri, Resident doctor in general surgery, Medical University of Vienna
Other Study IDs: 2049/2020
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient cohort:: all patients with vascular disorders consecutively admitted at our tertiary care hospital from March 16 to December 07, 2020
  Interventions: Diagnostic Test: PCR
- Control cohort:: data of two nationwide PCR-based studies conducted in a representative random sample, from April 1-6, and November 12-14, 2020, collected by the Austrian Ministry of Science and the Austrian Red Cross to estimate the spread of SARS-CoV-2 infection among the non-hospitalized Austrian population.
  Interventions: Diagnostic Test: PCR
- HCP cohort:: HCP worker data, including nurses, nurse technicians, physicians, surgical personal, physical therapists, nurse practitioners, environmental service workers, administrative staff, and dietitians, working in close proximity to admitted patients at our tertiary care hospital from March 16 to December 07, 2020.
  Interventions: Diagnostic Test: PCR

INTERVENTIONS:
Diagnostic Test: PCR — Nasal or pharyngeal respiratory swabs were routinely taken of each patient admitted at our departments and repeated regularly at 48 h intervals during the inpatient stay.
  In the HCP cohort testing for SARS-CoV-2 RNA was performed, on a weekly basis, at the Department of Laboratory Medicine, Medical University of Vienna, Austria, using real-time polymerase chain reaction (RT-PCR). Comparability of the results of all test methods used was confirmed by participation in international quality control ring trials.

SUMMARY:
Background: To investigate the prevalence of SARS-CoV-2 infection in hospitalized patients with vascular disorders after implementing institutional and governmental safety measures.

Materials and Methods: Vascular patients (VPs) admitted to our tertiary care hospital were routinely tested for SARS-CoV-2 infection on a two days basis between March and December, 2020. The prevalence of SARS-CoV-2 was compared between VPs and two independent Austrian populations (April and November 2020) tested by the Austrian Ministry of Science. The results were also compared to a cohort of health care personnel (HCP) working in close proximity to the study patients, tested weekly, between March and December, 2020. RT-PCR and antigen test were used to detect SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

All inpatient admissions

Exclusion Criteria:

Outpatient admissions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We investigated clinical data from all patients presenting at the hospital with vascular disorders, including peripheral artery disease (PAD), cardiac disorders (CD), aortic aneurysm (AA), extracranial artery disorders (EAD) and venous disorders (VD).
Sampling Method: Non-Probability Sample
Enrollment: 2243 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
prevalence of SARS-CoV-2 infection | March 16 to December 07, 2020
  The primary endpoint of the present study was to determine the prevalence of SARS-CoV-2 infection in patients with vascular disease after the implementation of institutional and governmental safety measures and compared it to SARS-CoV-2 infections among the general population in Austria.

CONTACTS AND LOCATIONS:
Overall Officials: Wolf W Eilenberg, MD. PhD., Study Chair — Wolf.eilenberg@meduniwien.ac.at
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
All study data will be made available upon request.